CLINICAL TRIAL: NCT02445235
Title: Study to Evaluate Outcomes of Patients Receiving Treatment for Wound Care, Pain Management or Surface Skin Scar Therapy
Acronym: SOPWS
Status: Terminated | Type: Observational
Why Stopped: Sponsor discretion determined no clinical benefit
Sponsor: Bracane Company (Industry)
Collaborators: IFG Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IFG2015-SOPWS
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Pain; Fungal Infection
Keywords: pain; wound care; fungal infections; scars; chronic pain; outcomes; PRO
MeSH Terms: conditions — Chronic Pain; Mycoses; Pain; Cicatrix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patient Reported Outcome Survey Tool — Patient Reported Outcome Survey Tool

SUMMARY:
This observational study is designed to evaluate the reported outcomes for patients receiving topical therapy for the treatment of pain, fungal infections or skin scars. The patients will complete the Patient Reported Outcome (PRO) survey monthly and provide valuable data on the patients perception of their health status and well being while receiving therapy.

DETAILED DESCRIPTION:
This observational study is designed to evaluate the reported outcomes for patients receiving topical therapy for the treatment of pain, fungal infections or skin scars. The patients will complete the Patient Reported Outcome (PRO) survey monthly and provide valuable data on the patients perception of their health status and well being while receiving therapy.

Patients are enrolled for 18 months. The investigator will complete a global patient assessment monthly of the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

1. An 18 to 85 years old (inclusive) female or male patient
2. Prescribed compound for the treatment of pain, wound healing or surface skin scar by their Principal Investigator
3. Any systemic disease (cardiac, renal, or hepatic) must be well controlled.
4. Has no skin lesions at the site of application of study medication except for wound under treatment
5. Able to provide informed consent

Exclusion Criteria:

1. Pregnant or lactating females or women at the child bearing potential not using effective contraception.
2. Use of other topical or transdermal medication. Patients may be withdrawn for a period of 2 weeks from all topical or transdermal medications prior to study initiation.
3. Hypersensitivity to local anesthetic or other ingredients of the compounded creams to be used in a study.
4. Prior reconstruction skin surgery or skin grafts in the area of cream application preventing absorption of cream except for the treatment of surface skin scar
5. Chronic pain conditions not expected to respond to topical pain medication such as deep abdominal pain, or from conditions such as cancer, or gouty arthritis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must be receiving therapy for pain, wound care or scar therapy
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Baseline PRO and Health Status Perception | Up to eighteen (18) months

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Nelson, RN, MS, Study Director — Bracane Company; Matt Fruge, BS, Study Chair — IFG Medical
Locations (3):
- United States (3):
  - BG Research, Lexington, Kentucky
  - Sevierville Foot and Ankle Clinic, Sevierville, Tennessee
  - Associates of Internal Medicine, Fort Worth, Texas